CLINICAL TRIAL: NCT00261417
Title: A Randomized, Double-Blind, Multicentre, Placebo-Controlled Study to Evaluate the Efficacy, Dose-Response and Safety of Tesaglitazar Therapy in Japanese Subjects With Type 2 Diabetes
Brief Title: Dose Response Study in Japanese Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The development program has been terminated
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D6160L00001; SH-SBD-0013
Record Dates: First submitted 2005-12-01; First posted 2005-12-05 (Estimated); Last update posted 2009-04-22 (Estimated); Status verified 2009-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — tesaglitazar

INTERVENTIONS:
Drug: Tesaglitazar

SUMMARY:
This is a 12-week study to determine the effect on glucose and lipids, safety, and tolerability of four doses of tesaglitazar (0.25, 0.5, 0.75 and 1 mg) compared with placebo in patients with type 2 diabetes. Improvement in dyslipidemia will be evaluated. The study comprises a 2-week screening period, 4-week placebo run-in, a 12-week randomized, double blind, parallel group, multi-center, placebo-controlled treatment period, and a 3-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Provision of a written informed consent
* Men or women who are >=18 years of age
* Female patients: postmenopausal, hysterectomized
* Diagnosed with type 2 diabetes
* Treated with diet alone or treatment with a single oral antidiabetic agent or low doses of two oral anti-diabetic agents

Exclusion Criteria:

* Type 1 diabetes
* New York Heart Association heart failure Class III or IV
* Treatment with chronic insulin
* History of hypersensitivity or intolerance to any peroxisome proliferator-activated receptor agonist (like Actos or Avandia), fenofibrate, metformin or 3-hydroxy-3-methylglutaryl coenzyme A reductase inhibitor (statin)
* History of drug-induced myopathy or drug-induced creatine kinase elevation, liver enzyme elevations, neutropenia (low white blood cells)
* Creatinine levels above twice the normal range
* Creatine kinase above 3 times the upper limit of normal
* Received any investigational product in other clinical studies within 12 weeks
* Any clinically significant abnormality identified on physical examination, laboratory tests or electrocardiogram, which in the judgment of the investigator would compromise the patient's safety or successful participation in the clinical study

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 2004-05; Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Dose-response relationship of tesaglitazar in subjects with type 2 diabetes by the assessment of the effects of each of four doses of tesaglitazar (0.25, 0.5, 0.75 and 1 mg) to placebo with respect to fasting plasma glucose

SECONDARY OUTCOMES:
Changes in the following variables from baseline to the end of the randomized treatment period:
Triglycerides, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol, very-low-density lipoprotein cholesterol, non-high-density lipoprotein cholesterol, total cholesterol apolipoproteins (Apo) (Apo A-I, Apo B and Apo CIII), and f
Glucose and insulin values during an oral glucose tolerance test
Effects on the reduction of insulin and glycosylated hemoglobin A1c levels
Effects on the proportion of fasting plasma glucose responders
Effects on the proportion of high-density lipoprotein cholesterol responders
Effects on the changes from baseline in weight and waist/hip ratio
Evaluate the pharmacokinetics of tesaglitazar
Assess the safety and tolerability of tesaglitazar compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Japan Medical Director, MD, Study Director — AstraZeneca
Locations (20):
- Japan (20):
  - Research Site, Ashino
  - Research Site, Fuchu Keijinkai
  - Research Site, Fujimino
  - Research Site, Hijirino Koike
  - Research Site, Houseikai
  - Research Site, Hyūga
  - Research Site, Iriuchijima
  - Research Site, Iwase
  - Research Site, Katō
  - Research Site, Kawamata
  - Research Site, Keishukai Shirakawa
  - Research Site, Koga
  - Research Site, Kōhoku
  - Research Site, Kōsei
  - Research Site, Kurosawa
  - Research Site, Nihonmatu
  - Research Site, Oki
  - Research Site, Saiseikai Fukuoka
  - Research Site, Sapporo
  - Research Site, Takamori